CLINICAL TRIAL: NCT00026338
Title: A Randomized Placebo Controlled Study Of OSI-774 (TARCEVA) Plus Gemcitabine In Patients With Locally Advanced, Unresectable Or Metastatic Pancreatic Cancer
Brief Title: Gemcitabine With/Out Erlotinib in Unresectable Locally Advanced/Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PA3; CAN-NCIC-PA3 (Other: PDQ); OSI-CAN-NCIC-PA3 (Other: OSI); CDR0000069020 (Other: PDQ)
Record Dates: First submitted 2001-11-09; First posted 2003-01-27 (Estimated); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Pancreatic Cancer
Keywords: stage III pancreatic cancer; adenocarcinoma of the pancreas; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Erlotinib Hydrochloride; Gemcitabine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- OSI-774 plus Gemcitabine (Active Comparator)
  Interventions: Drug: erlotinib hydrochloride; Drug: gemcitabine hydrochloride
- Placebo plus gemcitabine (Active Comparator)
  Interventions: Drug: gemcitabine hydrochloride

INTERVENTIONS:
Drug: erlotinib hydrochloride — 150 mg po daily
  Arms: OSI-774 plus Gemcitabine
Drug: gemcitabine hydrochloride — 1000 mg/m2 IV weekly (Cycle 1 -Day 1, 8, 15, 22, 29, 36, 43 of an 8 week cycle, Cycle 2 and subsequent cycles -Day 1,8 and 15 of a 4 week cycle)

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Biological therapies such as erlotinib use different ways to stimulate the immune system and stop cancer cells from growing. Combining chemotherapy and biological therapy may kill more tumor cells. It is not yet known if gemcitabine is more effective with or without erlotinib in treating pancreatic cancer.

PURPOSE: Randomized phase III trial to determine the effectiveness of gemcitabine with and without erlotinib in treating patients who have unresectable locally advanced or metastatic pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the overall survival rate in patients with unresectable locally advanced or metastatic pancreatic cancer treated with gemcitabine with or without erlotinib.
* Compare the progression-free survival rate in patients treated with these regimens.
* Compare the quality of life of patients treated with these regimens.
* Compare the response rate and response duration in patients treated with these regimens.
* Compare the nature, severity, and frequency of toxic effects of these regimens in these patients.
* Correlate the expression of tissue epidermal growth factor receptor levels at diagnosis with outcome and response in patients treated with these regimens.
* Determine the pharmacokinetics of erlotinib in these patients.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to participating center, extent of disease (locally advanced vs metastatic), and ECOG performance status (0-1 vs 2). Patients are randomized to one of two treatment arms.

* Arm I: Patients receive gemcitabine IV over 30 minutes on days 1, 8, 15, 22, 29, 36, and 43 of course 1 only, which lasts 8 weeks, and on days 1, 8, and 15 of all subsequent courses, which last 4 weeks each. Patients also receive 1 of 2 doses of oral erlotinib once daily.
* Arm II: Patients receive gemcitabine as in arm I and 1 of 2 doses of oral placebo once daily.

Treatment continues in both arms in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, on day 29 of course 1, on day 1 of all subsequent courses, at 4 weeks after study, and then every 12 weeks until disease progression.

Patients are followed at 4 weeks and then every 12 weeks thereafter.

PROJECTED ACCRUAL: A total of 800 patients (400 per treatment arm) will be accrued for this study within 11 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed adenocarcinoma of the pancreas
* Locally advanced or metastatic disease that is considered unresectable
* No known CNS metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Absolute granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin less than 2 times upper limit of normal (ULN)
* AST and/or ALT less than 2 times ULN (5 times ULN if liver metastases present)

Renal:

* Creatinine less than 1.5 times ULN

Cardiovascular:

* No uncontrolled high blood pressure
* No unstable angina
* No congestive heart failure
* No myocardial infarction within the past year
* No cardiac ventricular arrhythmias requiring medication

Gastrointestinal:

* No gastrointestinal (GI) tract disease resulting in an inability to take oral medication such as uncontrolled inflammatory GI disease (e.g., Crohn's disease or ulcerative colitis)
* No post-surgical malabsorption characterized by:

  * Uncontrolled diarrhea that results in weight loss and vitamin deficiency OR
  * Requires IV hyperalimentation
  * Pancreatic enzyme supplementation allowed provided that the above criteria are not met

Ophthalmic:

* No ocular inflammation or infection unless fully treated prior to study
* No significant ophthalmologic abnormalities, including the following:

  * Severe dry eye syndrome
  * Sjogren's syndrome
  * Keratoconjunctivitis sicca
  * Severe exposure keratopathy
  * Disorders that would increase the risk for epithelium-related complications (e.g., bullous keratopathy, aniridia, severe chemical burns, or neutrophilic keratitis)

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* No serious active infection
* No other serious underlying medical, psychological, or geographical condition that would preclude study participation
* No prior allergic reaction to compounds with similar chemical or biologic composition to erlotinib
* No other prior malignancy within the past 5 years except cancer in situ or basal cell or squamous cell skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent biologic therapy or immunotherapy

Chemotherapy:

* No prior chemotherapy except fluorouracil (with or without leucovorin calcium) or gemcitabine administered concurrently with radiotherapy as a radiosensitizer
* No other concurrent cytotoxic chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* See Chemotherapy
* At least 4 weeks since prior radiotherapy and recovered
* Prior radiotherapy for local disease allowed if evidence of disease progression has occurred
* No concurrent radiotherapy

Surgery:

* See Disease Characteristics
* At least 2 weeks since prior major surgery
* No concurrent ophthalmic surgery

Other:

* No prior epidermal growth factor receptor inhibitors
* At least 2 weeks since prior investigational drug
* No other concurrent investigational drugs during and for at least 30 days after study
* No other concurrent anti-cancer therapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 569 (Actual)
Dates: Start 2001-10-29 (Actual); Primary Completion 2004-09-17 (Actual); Study Completion 2009-02-10 (Actual)

PRIMARY OUTCOMES:
Overall survival | 3 years

SECONDARY OUTCOMES:
Progression free survival | 3 years
Quality of Life | 3 years
  Canada, US and selected countries only
Response rates | 3 years
  Complete and partial response only.
Toxicity | 3 years
EGFR levels | 3 years
  Correlate the expression oftissue EGFR levels (at diagnosis) with outcomes and response to treatment
Pharmacokinetics | 3 years
  To measure trough levels of081-774 (Tarceva™) to determine population pharmacokinetics

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm J. Moore, MD, Study Chair — Princess Margaret Hospital, Canada
Locations (173):
- United States (74):
  - Arizona Clinical Research Center, Tucson, Arizona
  - Highlands Oncology Group, Springdale, Arkansas
  - Alta Bates Comprehensive Cancer Center, Berkeley, California
  - Sutter Health West Cancer Research Group, Greenbrae, California
  - Loma Linda University Cancer Institute, Loma Linda, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Kenmar Research Institute, Los Angeles, California
  - Century City Hospital, Los Angeles, California
  - David Geffen School of Medicine, Los Angeles, California
  - Kaiser Permanente Medical Center/Kaiser Foundation Hospital - San Diego, San Diego, California
  - Davis, Posteraro, & Wasser, MDs, LLP, Manchester, Connecticut
  - New Britain General Hospital, New Britain, Connecticut
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - Hematology Oncology, P.C., Stamford, Connecticut
  - Florida Cancer Specialists, Fort Myers, Florida
  - Oncology-Hematology Group of South Florida, Miami, Florida
  - Ocala Oncology Center, Ocala, Florida
  - Oncology & Hematology Associates of West Broward, Tamarac, Florida
  - Moffitt Clinic at Tampa General Hospital, Tampa, Florida
  - Central Georgia Hematology Oncology, P.C., Macon, Georgia
  - Mountain States Tumor Institute, Boise, Idaho
  - Northwest Medical Specialists, P.C., Arlington Heights, Illinois
  - Veterans Affairs Medical Center - Hines (Hines Junior VA Hospital), Hines, Illinois
  - Oncology/Hematology Associates of Central Illinois, P.C., Peoria, Illinois
  - Midwest Cancer Research Group, Inc., Skokie, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Medical Consultants, Muncie, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Lucille Parker Markey Cancer Center, University of Kentucky, Lexington, Kentucky
  - Norton Healthcare Pavilion, Louisville, Kentucky
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Metairie, Louisiana
  - Tulane Cancer Center, New Orleans, Louisiana
  - Annapolis Medical Specialists, Annapolis, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Tuft-New England Medical Center, Boston, Massachusetts
  - St. Elizabeth's Medical Center, Boston, Massachusetts
  - Berkshire Physicians and Surgeons, P.C., Pittsfield, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Midwest Oncology Consortium, Kansas City, Missouri
  - New Hampshire Oncology-Hematology PA, Hooksett, New Hampshire
  - St. Barnabas Medical Center, Livingston, New Jersey
  - Hematology-Oncology Associates, Mount Holly, New Jersey
  - Cooper Cancer Institute, Voorhees Township, New Jersey
  - Cancer Center at Glens Falls Hospital, Glens Falls, New York
  - Arena Oncology Associates, Great Neck, New York
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - Beth Israel Medical Center, New York, New York
  - Interlakes Oncology/Hematology PC, Rochester, New York
  - Staten Island University Hospital, Staten Island, New York
  - University Hospital - Stony Brook, Stony Brook, New York
  - Presbyterian Hospital, Charlotte, North Carolina
  - Mid Dakota Clinic, P.C., Bismarck, North Dakota
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Earle A. Chiles Research Institute at Providence Portland Medical Center, Portland, Oregon
  - Hematology-Oncology Association of NE Pennsylvania, Dunmore, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Pennsylvania Oncology Hematology Associates, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Charleston Hematology-Oncology, P.A., Charleston, South Carolina
  - Sarah Cannon-Minnie Pearl Cancer Center, Nashville, Tennessee
  - Arlington Cancer Center, Arlington, Texas
  - Southwest Regional Cancer Center, Austin, Texas
  - Texas Cancer Care, Fort Worth, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Tyler Hematology Oncology, P.A., Tyler, Texas
  - Green Mountain Oncology Group, Bennington, Vermont
  - Hematology & Oncology Associates of Virginia, Mechanicsville, Virginia
  - Western Washington Oncology, Olympia, Washington
  - Southwest Washington Medical Center, Vancouver, Washington
  - Oncology of Wisconsin, Glendale, Wisconsin
- Argentina (7):
  - Hospital Britanico, Buenos Aires
  - Instituto de Oncologia Angel H. Roffo, Buenos Aires
  - Instituto Alexander Fleming, Buenos Aires
  - Hospital Churruca, Buenos Aires
  - Hospital Italiano, Buenos Aires
  - Hospital Interzonal De Augudos Euita, Lanús
  - Confidence Medical Center, San Isidro
- Australia (11):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Newcastle Mater Misericordiae Hospital, Newcastle, New South Wales
  - Institute of Oncology, Randwick, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Ashford Cancer Centre, Ashford, South Australia
  - Queen Elizabeth Hospital, Woodville, South Australia
  - Frankston Hospital, Frankston, Victoria
  - Austin and Repatriation Medical Centre, Heidelberg, Victoria
  - Royal Perth Hospital, Perth, Western Australia
  - Peter MacCallum Cancer Institute, Melbourne
- Institut Jules Bordet, Brussels, Belgium
- Brazil (3):
  - Nucleo de Oncologia da Bahia, Bahia
  - Hospital Santa Rita Irtmandade Santa Casa De Porto Alegre, Porto Alegre
  - Hospital Israelita Albert Einstein, São Paulo
- Canada (28):
  - Cross Cancer Institute, Edmonton, Alberta
  - British Columbia Cancer Agency - Centre for the Southern Interior, Kelowna, British Columbia
  - Penticton Regional Hospital, Penticton, British Columbia
  - British Columbia Cancer Agency - Fraser Valley Cancer Centre, Surrey, British Columbia
  - British Columbia Cancer Agency, Victoria, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Newfoundland Cancer Treatment and Research Foundation, St. John's, Newfoundland and Labrador
  - Queen Elizabeth II Health Science Centre, Halifax, Nova Scotia
  - Royal Victoria Hospital, Barrie, Barrie, Ontario
  - Cancer Care Ontario-Hamilton Regional Cancer Centre, Hamilton, Ontario
  - Kingston Regional Cancer Centre, Kingston, Ontario
  - Cancer Care Ontario-London Regional Cancer Centre, London, Ontario
  - Credit Valley Hospital, Mississauga, Ontario
  - Southlake Regional Health Centre, Newmarket, Ontario
  - Ottawa Regional Cancer Centre, Ottawa, Ontario
  - Peterborough Oncology Clinic, Peterborough, Ontario
  - Algoma District Medical Group, Sault Ste. Marie, Ontario
  - Hotel Dieu Health Sciences Hospital - Niagara, St. Catharines, Ontario
  - Toronto East General Hospital, Toronto, Ontario
  - Toronto Sunnybrook Regional Cancer Centre, Toronto, Ontario
  - Ontario Cancer Institute, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Saint Joseph's Health Centre - Toronto, Toronto, Ontario
  - Maisonneuve-Rosemont Hospital, Montreal, Quebec
  - Hopital Du Sacre-Coeur de Montreal, Montreal, Quebec
  - L'Hopital Laval, Ste-Foy, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
- Clinica Las Condes, Santiago, Chile
- China (2):
  - Pamela Youde Nethersole Eastern Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
- Germany (8):
  - Virchow Klinikum Humboldt Universitaet Berlin, Berlin
  - Universitaetsklinik und Strahlenklinik - Essen, Essen
  - Stadtische Kliniken Frankfurt-Hochst, Frankfurt
  - Tumor Biology Center at the Albert - Ludwigs University, Freiburg im Breisgau
  - Martin Luther Universitaet, Halle
  - Medizinische Universitaetsklinik und Poliklinik, Heidelberg
  - Universitatsklinik, Saarland, Homburg/Saar
  - University Wurzburg, Würzburg
- Greece (3):
  - University Hospital of Heraklion, Iraklion (Heraklion), Crete
  - Theagenio Medical Institute, Thessaloniki
  - Hippokration Hospital, Thessaloniki
- Prince of Wales Hospital, Shatin, New Territories, Hong Kong
- Israel (7):
  - Haemek Medical Center, Afula
  - Rambam Medical Center, Haifa
  - Rabin Medical Center - Beilinson Campus, Petah Tikva
  - Rabin Medical Center - Golda-Hasharon Campus, Petah Tikva
  - Kaplan Hospital, Rehovot
  - Tel-Aviv Sourasky Medical Center, Tel Aviv
  - Sheba Medical Center, Tel Litwinsky
- Policlinico - Cattedra di Ematologia, Palermo, Italy
- Mexico (2):
  - Instituto Nac de Cancerologia, Tlalpan, Mexico City
  - Centro Estatal de Cancerologia, Dviango
- New Zealand (2):
  - Auckland Hospital, Auckland
  - Christchurch Hospital, Christchurch
- Poland (2):
  - Great Poland Cancer Center, Poznan
  - Dolnoslaskie Centrum Oncology, Wroclaw
- Romania (4):
  - Institute of Oncology - Bucarest, Bucharest
  - Institutul Oncologic-Universitatea de Medicina, Cluj-Napoca
  - St. Spiridon University Hospital, Lasi
  - Clinical County Hospital of Sibiu, Sibiu
- Singapore (3):
  - National University Hospital, Singapore
  - Singapore General Hospital, Singapore
  - National Cancer Centre - Singapore, Singapore
- United Kingdom (13):
  - Queen Elizabeth Hospital, Birmingham, England
  - North Middlesex Hospital, Edmonton, London, England
  - St. Luke's Cancer Center, Guildford, England
  - Princess Royal Hospital, Hull, England
  - Saint Bartholomew's Hospital, London, England
  - Guy's and St. Thomas' Hospitals NHS Trust, London, England
  - Christie Hospital N.H.S. Trust, Manchester, England
  - Northern Centre for Cancer Treatment, Newcastle upon Tyne, England
  - Royal South Hants Hospital, Southampton, England
  - New Cross Hospital, Wolverhampton, England
  - Belfast City Hospital Trust, Belfast, Northern Ireland
  - Velindre Hospital, Cardiff, Wales
  - Churchill Hospital, Oxford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dhani NC, Tu D, Parulekar W, et al.: A retrospective analysis of tumor size (TS) as a continuous rather than discrete variable in advanced pancreatic cancer. [Abstract] J Clin Oncol 27 (Suppl 15): A-e15565, 2009.
- [Result] Moore MJ, da Cunha Santos G, Kamel-Reid S, et al.: The relationship of K-ras mutations and EGFR gene copy number to outcome in patients treated with Erlotinib on National Cancer Institute of Canada Clinical Trials Group trial study PA.3. [Abstract] J Clin Oncol 25 (Suppl 18): A-4521, 2007.
- [Result] Moore MJ, Goldstein D, Hamm J, Figer A, Hecht JR, Gallinger S, Au HJ, Murawa P, Walde D, Wolff RA, Campos D, Lim R, Ding K, Clark G, Voskoglou-Nomikos T, Ptasynski M, Parulekar W; National Cancer Institute of Canada Clinical Trials Group. Erlotinib plus gemcitabine compared with gemcitabine alone in patients with advanced pancreatic cancer: a phase III trial of the National Cancer Institute of Canada Clinical Trials Group. J Clin Oncol. 2007 May 20;25(15):1960-6. doi: 10.1200/JCO.2006.07.9525. Epub 2007 Apr 23. PMID 17452677
- [Result] Moore MJ, Goldstein D, Hamm J, et al.: Erlotinib improves survival when added to gemcitabine in patients with advanced pancreatic cancer. A phase III trial of the National Cancer Institute of Canada Clinical Trials Group [NCIC-CTG]. [Abstract] American Society of Clinical Oncology 2005 Gastrointestinal Cancers Symposium, 27-29 January 2005, Miami, Florida. A-77, 2005.